CLINICAL TRIAL: NCT05388552
Title: Clinical Features of Hyperkinetic Involuntary Movements Controlateral to Hemiplegia in Acute Stroke
Brief Title: Abnormal Hyperkinetic Movements Post Acute Stroke
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier de Saint-Denis (Other)
Responsible Party: Sponsor
Other Study IDs: CHSD_0018_NEURO; 2021-A03230-41 (Registry Identifier: IDRCB)
Record Dates: First submitted 2022-05-19; First posted 2022-05-24 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Neurology Department
Keywords: hyperkinetic movements; acute stroke
MeSH Terms: conditions — Hyperkinesis; Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The occurrence of abnormal movements is a frequent reason for consultation in neurology. The etiologies are broadly separated into "primary causes", intrinsically neurological diseases (of genetic or degenerative origin), and "secondary causes". In addition to certain medications or toxic substances, brain damage can be a cause. In this register, 22% of involuntary abnormal movements are related to a stroke and 1 to 4% of strokes are complicated by abnormal movements.

These are manifested by a parkinsonian syndrome or conversely by hypercinesia which can take the form of chorea or ballisms. Most hyperkinetic movements occur in the acute phase of the neurovascular event.

The frequency of these abnormal movements is still uncertain and their semeiological description has been the subject of only rare publications. It seems relevant to be interested in the frequency of these neurological phenomena and has their semeiologic characteristic

DETAILED DESCRIPTION:
The occurrence of abnormal movements is a frequent reason for consultation in neurology. The etiologies are broadly separated into "primary causes", in example intrinsically neurological diseases (of genetic or degenerative origin), and "secondary causes". In addition to certain medications or toxic substances, brain damage can be a cause. In this register, 22% of involuntary abnormal movements are related to a stroke and 1 to 4% of strokes are complicated by abnormal movements.

These are manifested by a parkinsonian syndrome or conversely by hypercinesia which can take the form of chorea or ballisms. Most hyperkinetic movements occur in the acute phase of the neurovascular event. . The pathophysiology seems simple and explained by a direct lesion or hypoperfusion of structures involved in the loops of the basal ganglia, especially when the putamen is affected. Intuitively, these abnormal hyperkinetic movements affect the contralateral hemibody to the vascular lesion, or the ipsilateral rating to the sensory and/ or motor deficit. However, observations have already been reported of involuntary hyperkinetic abnormal movements of the contralateral side to that presenting hemiplegia, i.e. in theorie controlled by a cerebral hemisphere free of acute cerebral lesion.

The frequency of these abnormal movements is still uncertain and their semeiological description has been the subject of only rare publications. A largest cohort reports abnormal involuntary movements very heterogeneous as to their clinical presentation (rotation of the head, orpharyngeal stereotypies to the limbs, compulsive manipulations of the environment or repeated passive mobilization of the contralateral limb paralyzed) In addition, the correlation of this type of neurological manifestations with vascular lesions has not yet been elucidated.

However, the unusual nature of this type of movement, it seems relevant to be interested in the frequency of these neurological phenomena and has their semeiologic characteristic.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age 18 years old)
* Patients with a stroke treated in the neurovascular intensive care unit of the Delafontaine Hospital in Saint-Denis (Hospitalization within 48 hours of the onset of the neurovascular episode
* Patients with abnormal hyperkinetic movements

Exclusion Criteria:

* Opposition of the patient or his entourage to participation in the registry
* Abnormal myoclonic movements of an epileptic nature
* Minor patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with abnormal hyperkinetic movements post-stroke, managed in the neurovascular intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2022-05-23 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
incidence of abnormal contralateral movements to hemiplegia in the acute phase of a stroke | Day 1
  incidence of abnormal contralateral movements to hemiplegia in the acute phase of a stroke

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital DELAFONTAINE, Saint-Denis, Île-de-France Region, France

REFERENCES:
- [Result] Mehanna R, Jankovic J. Movement disorders in cerebrovascular disease. Lancet Neurol. 2013 Jun;12(6):597-608. doi: 10.1016/S1474-4422(13)70057-7. Epub 2013 Apr 19. PMID 23602779
- [Result] Defebvre L, Krystkowiak P. Movement disorders and stroke. Rev Neurol (Paris). 2016 Aug-Sep;172(8-9):483-487. doi: 10.1016/j.neurol.2016.07.006. Epub 2016 Jul 28. PMID 27476417
- [Result] Vercueil L, Andriantseheno ML, Umeda Y, Carre S, Sellal F. Hyperkinesia contralateral to acute hemiplegia: relevance of previous frontal lesions. Parkinsonism Relat Disord. 2000 Apr 1;6(2):107-110. doi: 10.1016/s1353-8020(99)00059-0. PMID 10699392
- [Result] Ghika J, Bogousslavsky J, van Melle G, Regli F. Hyperkinetic motor behaviors contralateral to hemiplegia in acute stroke. Eur Neurol. 1995;35(1):27-32. doi: 10.1159/000117085. PMID 7737242